CLINICAL TRIAL: NCT05275582
Title: Developing a Team-Delivered Intervention for Smoking and Hazardous Drinking for Primary Care Veterans With Cardiovascular Diseases (CDA 18-006)
Brief Title: Developing a Team-Delivered Intervention for Smoking and Hazardous Drinking for Primary Care Veterans With Cardiovascular Diseases
Acronym: CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDX 22-006; CDA 18-006 (Other Grant/Funding Number: VA HSR&D); IK2HX002610 (NIH)
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Cigarette Use; Alcohol Use Above Recommended Limits; Cardiovascular Risk Factors (e.g., Hypertension); Cardiovascular Diseases
Keywords: Smoking; Drinking, alcohol; Cardiovascular diseases; Heart disease risk factors
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Smoking; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: The CARE intervention will be piloted in two formats: 1) that includes a conjoint meeting between a Patient Aligned Care Team (PACT) medical provider and a behavioral health provider; and 2) does not include the conjoint meeting with the medical provider. All other elements of the treatment are identical.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will not know which version of CARE that the patient receives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CARE-PACT (Experimental): Brief (5 minute) meeting between the PACT medical provider and a behavioral health educator (in person or virtual using VA's VA Video Connect (VVC) system) -followed by- 30 minute meeting alone with behavioral health educator (in person or virtual using VA's VVC system) 4 weeks of optional self monitoring using an app 2 optional 15-minute phone calls with behavioral health educator
  Interventions: Behavioral: CARE
- CARE-PCMHI (Experimental): 30 minute meeting alone with behavioral health educator (in person or virtual using VA's VVC system) 4 weeks of optional self monitoring using an app 2 optional 15-minute phone calls with behavioral health educator
  Interventions: Behavioral: CARE

INTERVENTIONS:
Behavioral: CARE — Behavioral intervention including
  -30 minute meeting alone with behavioral health educator (in person or virtual using VA's VVC system) 4 weeks of optional self monitoring using an app of substance use behavior, mood, other behavioral processes 2 optional 15-minute phone calls with behavioral health educator
  Other Names: CARE-PACT, CARE-PCMHI

SUMMARY:
In this study, the investigators are interested in learning how patients feel about and are impacted by a new approach for the primary care team to use to talk to patients about heart disease and health behaviors. The investigators were looking to recruit around 40 Veterans from Buffalo and Syracuse to be in this study. What it entailed is being randomly assigned to one of two conditions. If patients are assigned to the first condition, their upcoming primary care appointment will be extended by about 5 minutes because a Health Educator will join the end of that appointment. If they are assigned to the second condition they would have their typical primary care appointment. Beyond that, both conditions are quite similar. They will have an individual meeting following the primary care appointment with the Health Educator, two phone booster meetings at 2 and 4 weeks, and information about an optional app that they have the choice to use to help them track some health behaviors.

DETAILED DESCRIPTION:
Many Veterans (30.4%) with cardiovascular diseases (CVDs) continue to engage in behaviors that increase risk of cardiovascular events and early mortality, such as smoking or hazardous drinking. While the VA has several programs designed to help Veterans quit smoking or quit/reduce drinking, there is a gap in service for Veterans who are not ready for change-based treatments but continue to smoke or drink hazardously. VA Patient Aligned Care Teams (PACTs) screen all patients annually for alcohol and tobacco use, and thus the PACT platform is an ideal way to reach Veterans with CVDs who smoke and/or drink hazardously. Through the Primary Care Mental Health Integration (PCMHI) initiative, mental and behavioral health providers are embedded to provide effective, evidence-based, Veteran-centered, behavioral health interventions for a variety of co-occurring behavioral health concerns and medical problems. Educational and self-monitoring interventions are evidence-based and increase substance users' intentions to make a behavior change, and additionally improve patient factors including engagement, willingness to accept behavioral health referrals, and self-management strategies. This research proposal focuses on adapting elements of these evidence-based interventions specifically for a PACT-based VA setting to appeal to Veterans not yet ready to change smoking and/or drinking. This intervention aims to increase intention to change and may improve rates of cessation and engagement with change-based programs. The intervention will fill a gap in care and potentially improve the health and longevity of Veterans seen in PACT. The intervention, called CARE, will be piloted in two formats: 1) that includes a conjoint meeting between a PACT medical provider and a behavioral health provider; and 2) only with a behavioral health provider.

ELIGIBILITY:
Inclusion Criteria:

* Veteran patients age 18 seen in PACT at the Buffalo and Syracuse VA Medical Center (VAMCs) and catchment areas
* Upcoming PACT appointment
* A diagnosis of cardiac disease, including coronary artery disease, hypertension, hyperlipidemia, OR ischemia
* Positive alcohol or tobacco use screen for at least two consecutive years (including most recent) for:

  * a.Smoking (i.e., Answered "Yes" on the Annual Veteran's Health Administration (VHA) Tobacco Use Screening Questionnaire) AND/OR
  * b.Hazardous drinking (Alcohol Use Disorders-Consumption [AUD-C] 4 for men or 3 for women)
* Currently smokes at least one cigarette per day OR currently scores in a range indicating hazardous drinking on the Alcohol Use Disorders Identification Test (AUDIT) OR both [telephone screen]
* Currently reports on 1 to 10 scale having no greater than high-moderate (defined as 8) intention (i.e., 7) to change their drinking and/or smoking behavior [telephone screen]

Exclusion Criteria:

* Disorientation at time of eligibility (i.e., delirium, acute psychosis, dementia, severe intoxication) [from the electronic medical record (EMR), telephone screen, or clinical judgment at the time of the in person appointment]
* Unable to read or understand English [telephone screen]
* Non-Veteran status [EMR]

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Christina Gass, PhD, Principal Investigator — VA Western New York Healthcare System, Buffalo, NY
Locations (2):
- United States (2):
  - VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in May 2022 for the clinical trial and ended September of 2023. Veterans were identified via data pull/chart review for potential inclusion with inclusion criteria including having an upcoming primary care appointment, having a cardiovascular condition or risk factor, and screening positive on the last two annual tobacco use or alcohol use screens performed in primary care.
Groups:
- CARE-PACT: Brief (5 minute) meeting between the patient-aligned care team (PACT) medical provider and a behavioral health educator (in person or virtual using VA's Virtual Care (VVC) system) -followed by- 30 minute meeting alone with behavioral health educator (in person or virtual using VA's VVC system) 4 weeks of optional self monitoring using an app 2 optional 15-minute phone calls with behavioral health educator
  CARE: Behavioral intervention including
  -30 minute meeting alone with behavioral health educator (in person or virtual using VA's VVC system) 4 weeks of optional self monitoring using an app of substance use behavior, mood, other behavioral processes 2 optional 15-minute phone calls with behavioral health educator
- CARE-PCMHI: 30 minute meeting alone with behavioral health educator (in person or virtual using VA's VVC system) 4 weeks of optional self monitoring using an app 2 optional 15-minute phone calls with behavioral health educator
  CARE: Behavioral intervention including
  -30 minute meeting alone with behavioral health educator (in person or virtual using VA's VVC system) 4 weeks of optional self monitoring using an app of substance use behavior, mood, other behavioral processes 2 optional 15-minute phone calls with behavioral health educator
Period: Overall Study
Arm/Group | CARE-PACT | CARE-PCMHI
Started | 25 | 19
Completed | 18 | 17
Not Completed | 7 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Did not/could not complete primary care appointment for various reasons | 4 | 0
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- CARE-PACT: Brief (5 minute) meeting between the PACT medical provider and a behavioral health educator (in person or virtual using VA's VVC system) -followed by- 30 minute meeting alone with behavioral health educator (in person or virtual using VA's VVC system) 4 weeks of optional self monitoring using an app 2 optional 15-minute phone calls with behavioral health educator
  CARE: Behavioral intervention including
  -30 minute meeting alone with behavioral health educator (in person or virtual using VA's VVC system) 4 weeks of optional self monitoring using an app of substance use behavior, mood, other behavioral processes 2 optional 15-minute phone calls with behavioral health educator
- Total: Total of all reporting groups
Arm/Group | CARE-PACT | CARE-PCMHI | Total
Number analyzed (Participants) | 25 | 19 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (12.1) | 63.1 (14.1) | 62.7 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 24 | 19 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 18 | 14 | 32
  Race: Black | 6 | 5 | 11
  Race: Alaskan/Indigenous | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 19 | 44
Substance Targeted (Tobacco or Alcohol) [Count of Participants; unit: Participants]
  Tobacco | 16 | 12 | 28
  Alcohol | 9 | 7 | 16
Readiness to Change Drinking or Smoking [Mean (Standard Deviation); unit: units on a scale] — This is a 1-10 scale wherein participants are asked to rate their readiness to change drinking or smoking from 1-10 with 1 being not ready/not considering change up to 10, being taking steps toward change.
  This scale is based off of numerous "Readiness Rulers" published in the motivational interviewing literature.
  units on a scale | 5.0 (3.7) | 3.6 (2.9) | 4.4 (3.4)
Readiness to Change Questionnaire [Count of Participants; unit: Participants] — Readiness to Change Questionnaire. This is a standardized measure (Heather and Rollnick, 1993) with 12 items measuring how ready an individual is to make a change to a behavior (e.g., drinking, smoking). The scale contains subscales that can indicate which Stage of Change (Precontemplation, Contemplation, or Action) an individual is in during the time of measurement. It is scored by seeing which subscale an individual is highest on at the time of measurement (i.e., their highest subscale score among the three stages; if two subscale scores are equal then the higher stage is chosen).
  Participants
    Precontemplation | 5 | 6 | 11
    Contemplation | 13 | 10 | 23
    Action | 7 | 3 | 10
Cigarettes per Smoking Day [Mean (Standard Deviation); unit: cigarettes/smoking day] — This is one item from a two-item smoking quantity-frequency measure. Veterans were asked (1) on how many days of the last 28 did they smoke any cigarettes; and (2) on the days they smoked, how many they smoked. The second of those is reported here. The number corresponds directly to the average of how many cigarettes they smoked per smoking day in the past 28. 1=1 cigarettes per day, 2=2 cigarettes per day, etc. Population: Only those in the sample who were tobacco smokers were included in this analysis.
  cigarettes/smoking day
    number analyzed (Participants) | 16 | 12 | 28
    (all) | 10.1 (6.0) | 17.6 (12.7) | 12.9 (9.6)
Drinking Days [Mean (Standard Deviation); unit: Days] — This is one item from a two-item drinking quantity-frequency measure. Veterans were asked on how many days of the last 28 did they have at least one standard drink of alcohol. The number corresponds directly to the average of how many days they had a standard drink of alcohol in the past 28 days. 1=1 day out of 28 that they drank alcohol, 2=2 days per week that they drank alcohol, etc. Population: Only those who screened positive for alcohol use were included in this measure.
  Days
    number analyzed (Participants) | 9 | 7 | 16
    (all) | 21.2 (12.3) | 17.9 (9.8) | 19.8 (11.0)
Drinks per Drinking Day [Mean (Standard Deviation); unit: drinks/drinking day] — This is one item from a two-item drinking quantity-frequency measure. Veterans were asked (1) on how many days of the last 28 did they drink a standard drink of alcohol; and (2) on the days they drank, how many standard drinks they had. The second of those is reported here. The number corresponds directly to the average of how many drinks they consumed per drinking day in the past 28. 1=1 drink per drinking day, 2=2 drinks per drinking day, etc. Population: Only those who screened positive for alcohol use were included in this measure.
  drinks/drinking day
    number analyzed (Participants) | 9 | 7 | 16
    (all) | 4.1 (2.3) | 3.6 (2.2) | 3.9 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Readiness to Change Drinking OR Smoking
Description: Readiness to Change Questionnaire. This is a standardized measure (Heather and Rollnick, 1993) with 12 items measuring how ready an individual is to make a change to a behavior (e.g., drinking, smoking). The scale contains subscales that can indicate which Stage of Change (Precontemplation, Contemplation, or Action) an individual is in during the time of measurement. It is scored by seeing which subscale an individual is highest on at the time of measurement (i.e., their highest subscale score among the three stages; if two subscale scores are equal then the higher stage is chosen).
Time Frame: 6 weeks post intervention
Population: While the Baseline data include everyone who completed a baseline, this number reflects only those who continued in the study and received the intervention, and completed at least some outcome data (N=35). For this analysis, there are only 34, as one participant missed the 6 week assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | CARE-PACT | CARE-PCMHI
Number analyzed (Participants) | 17 | 17
Participants
  Precontemplation | 2 | 4
  Contemplation | 4 | 8
  Action | 11 | 5

2. Primary Outcome: Readiness to Change Drinking OR Smoking
Description: This is a 1-10 scale wherein participants are asked to rate their readiness to change drinking or smoking from 1-10 with 1 being not ready/not considering change up to 10, being taking steps toward change.
  This scale is based off of numerous "Readiness Rulers" published in the motivational interviewing literature.
Time Frame: 6 weeks post intervention
Population: While the Baseline data include everyone who completed a baseline, this number reflects only those who continued in the study and received the intervention, and completed at least some outcome data (N=35). For this analysis, there are only 34, as one participant missed the 6 week appointment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CARE-PACT | CARE-PCMHI
Number analyzed (Participants) | 17 | 17
units on a scale | 5.9 (3.4) | 4.6 (3.5)

3. Secondary Outcome: Cigarettes Per Day
Description: This is one item from a two-item smoking quantity-frequency measure. Veterans were asked (1) on how many days of the last 28 did they smoke any cigarettes; and (2) on the days they smoked, how many they smoked. The second of those is reported here. The number corresponds directly to the average of how many cigarettes they smoked per smoking day in the past 28. 1=1 cigarettes per day, 2=2 cigarettes per day, etc.
Time Frame: 6 weeks post intervention
Population: While the Baseline data include everyone who completed a baseline, this number reflects only those who continued in the study and received the intervention, and completed at least some outcome data (N=35). For this analysis, there are only 19 total, as one participant missed the 6 week appointment, and we only included those who smoked in the sample, and two who attended the 6-week appointment had missing data for this item.
Measure: Mean (Standard Deviation); unit: cigarettes/smoking day
Arm/Group | CARE-PACT | CARE-PCMHI
Number analyzed (Participants) | 8 | 11
cigarettes/smoking day | 6.4 (7.4) | 16.0 (16.6)

4. Secondary Outcome: Drinking Days
Description: This is one item from a two-item drinking quantity-frequency measure. Veterans were asked on how many days of the last 28 did they have at least one standard drink of alcohol. The number corresponds directly to the average of how many days they had a standard drink of alcohol in the past 28 days. 1=1 day out of 28 that they drank alcohol, 2=2 days per week that they drank alcohol, etc.
Time Frame: 6 weeks post intervention
Population: While the Baseline data include everyone who completed a baseline, this number reflects only those who continued in the study and received the intervention, and completed at least some outcome data (N=35). For this analysis, there are only 15 total, as one participant missed the 6 week appointment, and we only included those who smoked in the sample.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | CARE-PACT | CARE-PCMHI
Number analyzed (Participants) | 9 | 6
Days | 19.1 (12.0) | 22.3 (10.1)

5. Secondary Outcome: Drinks Per Drinking Day
Description: This is one item from a two-item drinking quantity-frequency measure. Veterans were asked (1) on how many days of the last 28 did they drink a standard drink of alcohol; and (2) on the days they drank, how many standard drinks they had. The second of those is reported here. The number corresponds directly to the average of how many drinks they consumed per drinking day in the past 28. 1=1 drink per drinking day, 2=2 drinks per drinking day, etc.
Time Frame: Six weeks post intervention
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: drinks/drinking day
Arm/Group | CARE-PACT | CARE-PCMHI
Number analyzed (Participants) | 9 | 6
drinks/drinking day | 3.4 (1.7) | 3.5 (2.3)

6. Secondary Outcome: Patient Satisfaction Survey
Description: This was a Patient Satisfaction Survey that assess for satisfaction with the healthcare system assessing satisfaction, quality, sense of care and concern, courtesy, and abilities of their providers.
  The scores reported are averages of the 7 items, with scores ranging from 1-5 with a 1 generally corresponding to poor and a 5 to excellent. One item is scaled as yes/maybe/no ("would you recommend the medical center to your friends/relatives) with a yes=5, maybe=3, and no=1.
Time Frame: 6 months post intervention
Population: While the Baseline data include everyone who completed a baseline, this number reflects only those who continued in the study and received the intervention, and completed at least some outcome data (N=35)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CARE-PACT | CARE-PCMHI
Number analyzed (Participants) | 18 | 17
units on a scale | 4.4 (0.7) | 3.8 (1.2)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the full period of data collection for the study (~2 years). For participants, they were monitored from their initial time in the study until their final assessment (~6 months).
Description: Serious Adverse Events were categorized as "related to study" or "unrelated to study" as determined by the respective Institutional Review Boards after review. "Unrelated to study" indicated that, while the serious adverse occurred during the study period, was determined by the review board to not be caused by or related to the study in any appreciable way.
Arm/Group | CARE-PACT | CARE-PCMHI
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/25 | 2/19
Other Adverse Events (participants affected / at risk) | 0/25 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CARE-PACT (N=25) | CARE-PCMHI (N=19)
Serious adverse event (Vascular disorders) | 0 (0) | 1 (1) — unrelated to study
serious adverse event (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — unrelated to study
Serious adverse event (General disorders) | 1 (1) | 0 (0) — unrelated to study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT05275582/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT05275582/ICF_000.pdf